CLINICAL TRIAL: NCT04785235
Title: The Effects of Non-Surgical Periodontal Therapy on Neutrophil Elastase and Elastase Alpha-1 Proteinase Inhibitor Levels in GCF in Periodontitis Patients With or Without Acute Coronary Syndrome
Brief Title: Neutrophil Elastase, Elastase Alpha-1 Proteinase, Periodontitis, Gingival Crevicular Fluid and Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Principal Investigator, Nilgün Özlem Alptekin, Clinical Professor, Baskent University
Other Study IDs: 05401018
Record Dates: First submitted 2021-02-09; First posted 2021-03-05 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Acute Coronary Syndrome; Periodontitis
MeSH Terms: conditions — Acute Coronary Syndrome; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — gingival crevicular fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ACS: Group ACS: Acute Coronary Syndrome
  Interventions: Procedure: Non-Surgical Periodontal Therapy
- Periodontitis: Group P :Periodontitis
  Interventions: Procedure: Non-Surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Therapy

SUMMARY:
Periodontitis may contribute to vascular damage, resulting in the destabilization of atherosclerotic plaque leading to acute coronary syndrome (ACS). In this study, we explored the effect of non-surgical periodontal treatment (NSPT) on cardiovascular blood biomarkers and gingival crevicular fluid (GCF) Neutrophil Elastase (NE) and α1-proteinase inhibitor (alpha-1PI) levels in periodontitis (P) participants with and without ACS.

Medical and dental examinations were performed to diagnose ACS and periodontitis, respectively. Seventeen patients with diagnosis ACS and periodontitis were included in this study, as a test group (Group ACS). Twenty-six, age and sex-matched control patients with periodontitis (Group P) were otherwise systemically healthy. Both groups received NSPT. Plasma levels of cholesterol, triglyceride, high-density lipoprotein (HDL), low-density lipoprotein (LDL), C-reactive protein (CRP), GCF NE activity, and GCF α1-PI levels were measured baseline, at1st and 3rd months after NSPT.

DETAILED DESCRIPTION:
This research was approved by the human participants ethics board of Selcuk University Faculty of Dentistry (project number=301) and was conducted in accordance with the Helsinki Declaration of 1975, as revised in 2013. Informed consent was obtained from patients prior to oral diagnostic examination.

Inclusion criteria for ACS group :

• Patients diagnosed with both ACS and localized or generalized periodontitis of stage II or III with grade B or C.

The diagnosis of ACS was performed by a consultant cardiologist based on clinical signs and symptoms of cardiac ischemia, cardiac enzyme levels, changes in electrocardiography, and results of echocardiography and coronary angiography, according to the guidelines of American College of Cardiology/American Heart Association . The test group of ACS patients myocardial infarction (NSTEMI), and ST-segment elevation myocardial infarction (STEMI) were hospitalized in Selcuk University Meram Medical Faculty Department of Cardiology (Konya/Turkey).Unstable angina (UA) was defined as the new onset or a changed pattern of angina over the past 2 months and Canadian Cardiovascular Society (CCS) class IV angina at the time of presentation coinciding with appropriate objective evidence of myocardial ischemia on an electrocardiogram (ECG) or myocardial perfusion imaging. ACS with ST-segment elevation was defined as AMI characterized by: chest pain, radiating or not to the upper extremities, lower jaw, upper back or epigastrium lasting 30 minutes or more, associated or not with sweating, nausea or pallor; presence of ST-segment elevation of 1 mm in two or more contiguous peripheral leads or 2 mm in two or more contiguous precordial leads on electrocardiogram (ECG); and elevation in serum markers of myocardial injury and necrosis (CK, CK-MB) three times their reference value28. Non-ST-segment elevation ACS on ECG was defined as a clinical condition similar to that mentioned above but with chest pain lasting less than 30 minutes, with or without elevation of serum enzyme markers of myocardial injury and necrosis (CK, CK-MB, cardiac troponins I and T). ACS patients were referred to the Department of Periodontology, Faculty of Dentistry, Selcuk University (Konya/Turkey) for periodontal examination in a one- year period.

Inclusion criteria for control group :

• Patients diagnosed with localized or generalized periodontitis of stage II or III with grade B or C.

Exclusions for both groups included

* metabolic disorders,
* high blood pressure,
* treated with antihypertensive medications,
* periodontal therapy antibiotic treatment until 3 months prior the study. Smoking habits and education status were also recorded. ACS patients take aspirin (1 × 100 mg per day) during 1 month.This study was supported by grants from the Selcuk University Scientific Research Projects (05401018).

Clinical Periodontal Examination All surviving individuals with ACS underwent a thorough periodontal examination approximately 1 month after treatment and hospital release. All participants were evaluated for oral health clinically and radiographically. The periodontal condition was graded based on the current classification method for periodontal diseases and subjects with localized or generalized periodontitis of stage II or III with grade B or C were selected. Periodontal health status of patients was evaluated by plaque index (PI), papilla bleeding index , probing depth (PD) and clinical attachment level (CAL). All probing scores were measured with Williams periodontal probe calibrated in millimeters. Clinical attachment loss was determined relative to the cementoenamel junction. Periodontal index was evaluated for risk of infectiousness (PIRI) scores.

Gingival Crevicular Fluid Samples:

At baseline, GCF samples were collected for each subject from 4 distinct inter-proximal sites (one site for each quadrant). Sampling sites were chosen only at the buccal directions of the inter-proximal regions of molar teeth with PD more than 5 mm. The four GCF samples for each subject in the two research groups were pooled to ensure sufficient sensitivity for each subject. Consequently, site-specific differences were not evaluated. The same sites were sampled at 1 and 3 months following treatment. Sites were isolated with cotton rolls, gently dried with air syringe and the obvious supra-gingival plaque was carefully removed with a curette. GCF was collected with prefabricated paper strips . The strip was inserted into the pocket until mild resistance was felt and kept there for 30 seconds. Contaminated samples with blood or saliva were discharged. The volume of GCF was determined with Periotron 8000 previously calibrated with serum . Four strips were pooled in a single tube containing 500microliter phosphate buffered saline (PBS), pH 7.4 and, repeated, for each patient. The tubes were vortexed for 10 min and stored at -80 C until assayed.

ELIGIBILITY:
Inclusion criteria for ACS group :

• Patients diagnosed with both ACS and localized or generalized periodontitis of stage II or III with grade B or C. ACS patients myocardial infarction (NSTEMI), and ST-segment elevation myocardial infarction (STEMI) were hospitalized .

Unstable angina (UA) was defined as the new onset or a changed pattern of angina over the past 2 months and Canadian Cardiovascular Society (CCS) class IV angina at the time of presentation coinciding with appropriate objective evidence of myocardial ischemia on an electrocardiogram (ECG) or myocardial perfusion imaging. ACS with ST-segment elevation was defined as AMI characterized by: chest pain, radiating or not to the upper extremities, lower jaw, upper back or epigastrium lasting 30 minutes or more, associated or not with sweating, nausea or pallor; presence of ST-segment elevation of 1 mm in two or more contiguous peripheral leads or 2 mm in two or more contiguous precordial leads on electrocardiogram (ECG); and elevation in serum markers of myocardial injury and necrosis (CK, CK-MB) three times their reference value28. Non-ST-segment elevation ACS on ECG was defined as a clinical condition similar to that mentioned above but with chest pain lasting less than 30 minutes, with or without elevation of serum enzyme markers of myocardial injury and necrosis (CK, CK-MB, cardiac troponins I and T). ACS patients were referred to the Department of Periodontology, Faculty of Dentistry, Selcuk University (Konya/Turkey) for periodontal examination in a one- year period.

Inclusion criteria for control group :

• Patients diagnosed with localized or generalized periodontitis of stage II or III with grade B or C.

Twenty-six age and sex-matched patients (43.04±8.35 years) with periodontitis (Group P) otherwise systemically healthy were recruited as control group in the Department of Periodontology, Faculty of Dentistry, Selcuk University (Konya/Turkey).

Exclusions for both groups included

* metabolic disorders,
* high blood pressure,
* treated with antihypertensive medications,
* periodontal therapy antibiotic treatment until 3 months prior the study. Smoking habits and education status were also recorded. ACS patients take aspirin (1 × 100 mg per day) during 1 month.

Ages: 35 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: The periodontal condition was graded based on the current classification method for periodontal diseases and subjects with localized or generalized periodontitis of stage II or III with grade B or C were selected
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2007-10-15 (Actual); Primary Completion 2008-10-15 (Actual); Study Completion 2008-10-15 (Actual)

PRIMARY OUTCOMES:
GCF NE levels | in 3months
  Change of NE levels in ACS patients after NSPT.
GCF α1-PI | in 3months
  Change of GCF α1-PI in ACS patients after NSPT.

SECONDARY OUTCOMES:
change in NE / α1-PI rates | in 3months
  Change of in NE / α1-PI rates in ACS patients after NSPT.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Ozlem Alptekin, prof.dr, Study Director — Baskent Univercity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liljestrand JM, Paju S, Pietiainen M, Buhlin K, Persson GR, Nieminen MS, Sinisalo J, Mantyla P, Pussinen PJ. Immunologic burden links periodontitis to acute coronary syndrome. Atherosclerosis. 2018 Jan;268:177-184. doi: 10.1016/j.atherosclerosis.2017.12.007. Epub 2017 Dec 6. PMID 29232563
- [Background] Bokhari SA, Khan AA, Butt AK, Azhar M, Hanif M, Izhar M, Tatakis DN. Non-surgical periodontal therapy reduces coronary heart disease risk markers: a randomized controlled trial. J Clin Periodontol. 2012 Nov;39(11):1065-74. doi: 10.1111/j.1600-051X.2012.01942.x. Epub 2012 Sep 11. PMID 22966824
- [Background] Montenegro MM, Ribeiro IWJ, Kampits C, Saffi MAL, Furtado MV, Polanczyk CA, Haas AN, Rosing CK. Randomized controlled trial of the effect of periodontal treatment on cardiovascular risk biomarkers in patients with stable coronary artery disease: Preliminary findings of 3 months. J Clin Periodontol. 2019 Mar;46(3):321-331. doi: 10.1111/jcpe.13085. Epub 2019 Mar 6. PMID 30761568
- [Derived] Ye Z, Cao Y, Miao C, Liu W, Dong L, Lv Z, Iheozor-Ejiofor Z, Li C. Periodontal therapy for primary or secondary prevention of cardiovascular disease in people with periodontitis. Cochrane Database Syst Rev. 2022 Oct 4;10(10):CD009197. doi: 10.1002/14651858.CD009197.pub5. PMID 36194420
- [Derived] Kayar NA, Ustun K, Gozlu M, Haliloglu S, Alptekin NO. The effects of non-surgical periodontal therapy on neutrophil elastase and elastase alpha-1 proteinase inhibitor levels in GCF in periodontitis patients with or without acute coronary syndrome. Clin Oral Investig. 2021 May;25(5):3329-3338. doi: 10.1007/s00784-021-03838-3. Epub 2021 Mar 9. PMID 33687554